CLINICAL TRIAL: NCT05377216
Title: Characterization of Cardiac Electrophysiological Effects of Autonomic Neuromodulation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 851066
Record Dates: First submitted 2022-05-02; First posted 2022-05-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stellate ganglion block (Experimental): All subjects will undergo stellate ganglion block during their VT ablation procedure
  Interventions: Drug: Stellate Ganglion Block

INTERVENTIONS:
Drug: Stellate Ganglion Block — Left sided percutaneous stellate ganglion block

SUMMARY:
Prospective cohort study evaluating the electrophysiologic and biochemical effects of stellate ganglion block in patients with ventricular tachycardia.

ELIGIBILITY:
Inclusion Criteria:

* Planned catheter based VT ablation
* Age at least 18 years

Exclusion Criteria:

* Pregnancy
* Contraindication to SGB or VT ablation
* Hypersensitivity of local anesthetic of amide type
* Hemodynamic instability during the procedure prior to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Ventricular Effective Refractory Period | 30 minutes following stellate ganglion block
  Change in Ventricular Effective Refractory Period at 600ms drive train (measured in milliseconds)

SECONDARY OUTCOMES:
Ventricular Arrhythmia Inducibility | 30 minutes following stellate ganglion block
  Induction of monomorphic ventricular arrhythmia (binary outcome) during ventricular programmed stimulation
Neuropeptide Y | 30 minutes following stellate ganglion block
  Change in level of neuropeptide Y from baseline (measured in pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided